CLINICAL TRIAL: NCT01699022
Title: Pharmacokinetic and Pharmacodynamic Study of Cyclofem
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A09-109
Record Dates: First submitted 2012-09-28; First posted 2012-10-03 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Contraception
Keywords: Contraceptive; Injectable
MeSH Terms: interventions — CycloProvera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection Cyclofem (Experimental): Injection of Cyclofem contains 25 mg medroxyprogesterone acetate (MPA) and 5 mg estradiol cypionate as a microcrystalline suspension in 0.5ml aqueous solution and is supplied in vials.
  Women were administered three consecutive monthly injections of Cyclofem for prevention of ovulation, and were followed until the 92nd day from the last (third) injection.
  Interventions: Drug: Injection Cyclofem

INTERVENTIONS:
Drug: Injection Cyclofem — Injection Cyclofem contains 25 mg medroxyprogesterone acetate (MPA) and 5 mg estradiol cypionate as a microcrystalline suspension in 0.5ml aqueous solution and is supplied in vials.
  Women were administered three consecutive monthly injections of Cyclofem for prevention of ovulation, and were followed until the 92nd day from the last (third) injection.
  Other Names: Cyclofem

SUMMARY:
Cyclofem® is a monthly injectable contraceptive containing 25 mg of medroxyprogesterone acetate (MPA) and 5 mg of estradiol cypionate (E2C), a long-acting ester of estradiol. The current study will assess the steady-state pharmacokinetics and pharmacodynamics of medroxyprogesterone acetate (MPA) and estradiol (E2) after administration of Cyclofem® and will provide critical information to determine similar bioavailability of Cyclofem to Lunelle in women residing in the United States of America.

DETAILED DESCRIPTION:
Concept Foundation, an international nonprofit organization based in Bangkok, Thailand, was given the commercial rights to Cyclofem® by the World Health Organization (WHO) for use internationally. The brand names that the Concept Foundation has registered internationally include Cyclofem®, and Novafem® (Pharmacia Pharmaceuticals, Peapack NJ, formerly (Pharmacia and Upjohn of Kalamazoo, Michigan). The company launched its product under license from Concept Foundation with their own brand name, Lunelle™ in the US market. Lunelle™ was approved by the Food and Drug Administration (FDA) in October, 2000 following which approximately 350,000 women had used the product. However, following the acquisition of Pharmacia and Upjohn by Pfizer and due to several production problems, Pfizer withdrew Lunelle™ from the United States (US) market. Concept Foundation has licensed Sun Pharmaceutical Industries Ltd, Mumbai, India to manufacture and market Cyclofem® in India and other developing countries. United States Food and Drug Administration (US FDA) approval of Cyclofem® is pivotal to the ultimate acceptance of such products in many countries because of the rigorous standards applied by the Food and Drug Administration (FDA) for drug safety and efficacy. This initial pharmacokinetic (PK) study is the first step on the road to Food and Drug Administration (FDA) approval with the ultimate goal to expand the access and range of methods available to women in the public sector. Approval of Cyclofem® by the United States Food and Drug Administration (US FDA) would also allow the reintroduction of CICs to the United States (US) market.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 45 years of age, inclusive;
2. In good health, as evidenced by history and procedures at screening/enrollment visit
3. Without any clinically significant systemic disease;
4. Not at risk for pregnancy, having undergone surgical sterilization
5. Have had regular menstrual cycles (every 21-35 days) for the past two cycles;
6. Planning to reside in the area for at least 7 months after enrolling in the study; and
7. Willing and able to comply with study procedures
8. Have a body mass index (BMI) between 18 and 30 inclusive.

Exclusion Criteria:

1. Contraindications to the use of Cyclofem® include:

   1. Smoking any number of cigarettes per day in a woman > 35 years old (or in a woman 34 years-old who will turn 35 years-old during the study),
   2. Symptoms of chest pain or shortness of breath,
   3. Screening visit blood pressure >140/90, (subjects on hypertensive medications, in good blood pressure control will be admitted).
   4. Past or current thrombophlebitis or thromboembolic disorders,
   5. Past or current cerebral vascular or coronary artery disease
   6. History of stroke, myocardial infarction or ischemic heart disease or complicated valvular heart disease
   7. Diabetes
   8. Past or current carcinoma of the endometrium cervix or vagina; breast or other known or suspected estrogen-depended neoplasia,
   9. Headaches with focal neurological symptoms,
   10. Unexplained abnormal vaginal bleeding,
   11. Liver dysfunction or disease, such as a history of hepatic adenoma or carcinoma; history of cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use including severe pruritus of pregnancy, severe cirrhosis, or active hepatitis (defined as aspartate aminotransferase [AST or SGOT ≥ 120 IU/L] or alanine aminotransferase [ALT or SGPT ≥ 135 IU/L]) or clinically significant laboratory abnormalities as judged by the physician evaluating the individual subject).
2. Known hypersensitivity to any component of Cyclofem®
3. Have an abnormal Pap smear in the past 12 months defined as:

   1. Atypical squamous cells of undetermined significance (ASC-US) without a normal repeat Pap smear at least 6 months later;
   2. Atypical squamous cells of undetermined significance (ASC-US) with positive reflex high-risk human papillomavirus (HPV) testing (Atypical squamous cells of undetermined significance [ASC-US]/human papillomavirus [HPV]+) or low-grade squamous intraepithelial lesion (LSIL) except when a colposcopy was performed (with or without biopsy) and found no evidence of high-grade disease (cervical intraepithelial neoplasia [CIN II] or worse) unless treatment is indicated per local standard of care;
   3. ASC-H, atypical glandular cells, or high grade squamous intraepithelial lesion (HSIL) unless treatment was received and follow-up at least 6 months after the treatment showed no evidence of disease; malignant cells;
4. Current use of rifampin, griseofulvin, phenytoin, carbamazepine, barbiturates, or primidone;
5. Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol, such as any major chronic illness including cancer, serious autoimmune disease or a major psychiatric disorder (e.g. schizophrenia);
6. Current participation in any other drug or device study, or any study which, in the opinion of the investigator, would jeopardize interpretation of results of this study;
7. Active thyroid disease as measured by thyroid-stimulating hormone [TSH] levels ≤0.3 mU/L or ≥ 5 mU/L. Subjects with thyroid disease in good control with thyroid medication will be admitted.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Principal Investigator — Director, Conrad Clinical Research Center.
Locations (1):
- Clinical Research Center Norfolk, Virginia 601 Colley Avenue,, Norfolk, Virginia, United States

REFERENCES:
- [Derived] Thurman A, Kimble T, Hall P, Schwartz JL, Archer DF. Medroxyprogesterone acetate and estradiol cypionate injectable suspension (Cyclofem) monthly contraceptive injection: steady-state pharmacokinetics. Contraception. 2013 Jun;87(6):738-43. doi: 10.1016/j.contraception.2012.11.010. Epub 2012 Dec 22. PMID 23265980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the CONRAD Clinical Research Center (CRC) located in the Jones Institute for Reproductive Medicine at the Eastern Virginia Medical School (EVMS) in Norfolk, vasectomy (VA) in subjects with previous surgical sterilization and therefore were not at risk for pregnancy
Pre-assignment Details: A total of 7 women failed screening: 3 women had control cycle luteal phase serum P < 3 ng/mL; 3 women withdrew consent; and 1 potential subject was not enrolled because the study had enrolled the requisite number of subjects and was closed for enrollment
Period: Overall Study
Arm/Group | Injection Cyclofem
Started | 17
Completed | 14
Not Completed | 3
Not completed — Early discontinuation from the study | 3

BASELINE CHARACTERISTICS:
Arm/Group | Injection Cyclofem
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (5.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Medroxyprogesterone Acetate (MPA) Concentrations
Description: Assessment of mean trough levels of medroxyprogesterone acetate (MPA) on Day 1, Day 29, Day 57 and Day 85
Time Frame: "Day 1", "Day 29", "Day 57' and 'Day 85"
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Injection Cyclofem
Number analyzed (Participants) | 17
ng/mL
  Day 1 | 0.00 (0.02)
  Day 29 | 0.27 (0.09)
  Day 57 | 0.43 (0.13)
  Day 85 | 0.44 (0.19)

2. Primary Outcome: Medroxyprogesterone Acetate (MPA) Pharmacokinetics
Description: The mean serum concentration-time profile for medroxyprogesterone acetate (MPA) after three consecutive monthly intramuscular administration of Cyclofem (AUC). Peripheral blood sample for MPA was to be drawn three times a week for PK assessment during the third treatment month (Days 58, 60, 62, 64, 67, 69, 71, 75, 78, and 85) and for Day 85 (28 days post 3rd dose).
Time Frame: "Day 85"
Measure: Mean (Standard Error); unit: ng*day/mL
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
ng*day/mL
  AUC (0-84) | 31.5029 (7.49456)
  AUC (0-28) | 20.5831 (6.58448)
  AUC (0-inf) | 33.4528 (8.23617)

3. Primary Outcome: Medroxyprogesterone Acetate (MPA) Pharmacokinetics Cmax
Description: The mean serum concentration-time profile for medroxyprogesterone acetate (MPA) after three consecutive monthly intramuscular administration of Cyclofem
Time Frame: 85 days
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
ng/mL | 1.311380 (0.437259)

4. Primary Outcome: Medroxyprogesterone Acetate (MPA) Pharmacokinetics Tmax
Description: Mean serum medroxyprogesterone acetate (MPA) concentrations peaked at 4.1 days (range 1 - 21 days) after the third monthly administration of Cyclofem.
Time Frame: "Day 85"
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Cyclofem
Number analyzed (Participants) | 15
day | 4.1 (5.01)

5. Primary Outcome: Medroxyprogesterone Acetate (MPA) Pharmacokinetics T1/2
Time Frame: "Day 85"
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
day | 16.9413 (7.49264)

6. Primary Outcome: Estradiol (E2) Concentrations
Description: Mean serum estradiol (E2) concentrations on Day 1, Day 29, Day 57 and Day 85
Time Frame: "Day 1", "Day 29", "Day 57' and ''Day 85"
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
pg/mL
  Day 1 | 46 (18)
  Day 29 | 44 (19)
  Day 57 | 52 (22)
  Day 85 | 42 (17)

7. Primary Outcome: Estradiol (E2) Pharmacokinetics.
Description: AUC 0-28, AUC(0-inf). Peripheral blood sample for E2 was to be drawn three times a week for PK assessment during the third treatment month.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: pg*day/mL
Arm/Group | Injection Cyclofem
Number analyzed (Participants) | 17
pg*day/mL
  AUC (0-28) | 3289.6546 (888.56879)
  AUC (0-inf) | 3922.3365 (1019.80283)

8. Primary Outcome: Tmax
Description: Mean serum concentrations of estradiol (E2) peaked by 3.3 days (range 1 - 7 days) following the third monthly injection
Time Frame: "Day 85"
Population: Tmax
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
day | 3.3 (2.49)

9. Primary Outcome: T1/2
Description: Mean no of days for medroxyprogesterone acetate (MPA) and estradiol (E2)
Time Frame: "Day 85"
Population: Tmax
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
day
  medroxyprogesterone acetate (MPA) | 16.9413 (7.49264)
  Estradiol (E2) | 10.0960 (4.87120)

10. Primary Outcome: Number of Participants Who Achieved Ovulation Determined by Serum Progesterone Concentration
Description: Return of ovulation measured by changes in serum progesterone concentration by
  analysis on Day 18, Day 21 (Control cycle), Day 103, Day 106, Day 131 and Day 134 indicating the number of subjects who achieved ovulation.
  Outcome measure description indicates what was measure.
Time Frame: Day 134
Measure: Number; unit: participants
Arm/Group | Cyclofem
Number analyzed (Participants) | 17
participants
  Day 18 | 17
  Day 21 | 17
  Day 103 | 0
  Day 106 | 1
  Day 131 | 1
  Day 134 | 1

ADVERSE EVENTS:
Time Frame: The subjects were assessed for incidence of adverse events up to Day 92 (during the control and treatment period, and up to Day 134 (during the follow-up period)
Description: Toxicities and AEs were summarized by severity and relationship to treatment. Clinical laboratory parameters and vital signs were summarized as changes and shifts from baseline to final on treatment assignment and by clinically significant abnormalities. Vital signs during study drug dosing were summarized as changes from baseline.
Arm/Group | Injection Cyclofem
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 7/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injection Cyclofem (N=17)
Menorrhagia (Reproductive system and breast disorders) | 7 (7)
Vaginitis bacterial (Infections and infestations) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No